CLINICAL TRIAL: NCT04257942
Title: Pathological Crystallization of Cholesterol in Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Dr. Chen Speter, doctor, Sheba Medical Center
Other Study IDs: SHEBA - 19 - 6467 - MH - CTIL
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Crystallization of Cholesterol in Atherosclerosis
MeSH Terms: interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — atheromas that are being removed from arteries
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: carotid endarterectomy — carotid endarterctomy that is being used for carotid stenosis disease

SUMMARY:
Endarterectomy of the carotid artery procedure will be performed at Sheba Medical center vascular surgery department, followed by fixation and histology. Tissues will then be transferred to Weizmann Institute of Science for observation implementing advanced electron microscopy techniques. Finally, joint evaluation of the results will be carried out, in relation to the patient clinical history.

DETAILED DESCRIPTION:
Human atherosclerotic tissues will be obtained from the Department of Vascular Surgery, Sheba Medical Center. Tissues will be taken from donors undergoing routine endarterectomy procedures.We chose carotid artery as the source for the atheromas, due to its high prevalence and its considerable size.All speciemnts will be studied in Cryo-Scanning Electron Microscopy (Cryo-SEM). Tissues will be observed in hydrated vitrified state, after High Pressure Freezing (HPF) and freeze fracture, as well established in the WIS group. Samples will be observed at -120°C. Cathode-Luminescence (CL) detects a luminescence signal induced by electrons in cholesterol crystals and CE condensed states. It will be implemented herein under cryogenic conditions. Sample preparation is as for cryo-SEM. Cryo-FIB-SEM block face serial imaging allows the acquisition of serial images over large volumes (tens of cubed micrometers), at a relatively high imaging resolution (up to 5nm3 voxel size). Volumes of up to 40x40x40 ml will be imaged with a resolution of up to 10nm. The data will be minimally processed and aligned using FIJI, reconstructed and manually segmented using Avizo Lite 9.2.0 software.

ELIGIBILITY:
Inclusion Criteria:

* all patients that are being operated on for carotid endarterctomy due to carotid stenosis

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with carotid stenosis - symptomatic and asymptomatic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
crystallization of cholesterol in atherosclerosis | 3 years
  Understand the interrelation between structural, morphological and spatial characteristics of cholesterol crystals found within the atherosclerotic lesion and its maturation and destabilization.

IPD SHARING:
Plan to Share IPD: Yes
only the pthological and clinical findings
Supporting Information: Study Protocol, ICF
Time Frame: 2023- forever